CLINICAL TRIAL: NCT00966550
Title: Tomato Products and Postprandial Oxidation and Inflammation: a Clinical Trial in Healthy Weight Men and Women
Brief Title: A Study of Tomato Products and Disease Risk
Acronym: TOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Collaborators: Tomato Products Wellness Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: TOM 2009-071
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Results first posted 2014-10-16 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-02

CONDITIONS: Inflammation
Keywords: Tomato; Nutrition
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tomato (Active Comparator): Tomato with high carb/fat meal
  Interventions: Other: Tomato
- Non-Tomato (Placebo Comparator): Non-tomato with high carb/fat meal
  Interventions: Other: Non-tomato

INTERVENTIONS:
Other: Tomato — Tomato with high carb/fat meal
  Other Names: Active Comparator
  Arms: Tomato
Other: Non-tomato — Non-tomato with high carb/fat meal
  Other Names: Placebo Comparator
  Arms: Non-Tomato

SUMMARY:
The purpose of this research study is to test whether certain compounds in tomatoes will help reduce factors in the subject's blood associated with disease risk. The investigators want to know if the tomato-associated compounds will lower or improve the status of these factors, like cholesterol and inflammation. In this research study, the subject will be asked to consume high fat test meals on two separate occasions. The investigators want to see how the subject's body responds to a standard high fat meal, one meal with tomato products and one meal without tomato products. The investigators will measure the subject's blood throughout the study period to determine if consumption of tomato products reduces factors in their blood associated with disease risk.

DETAILED DESCRIPTION:
This study will take three weeks at most, and require one initial screening visit lasting approximately 45 minutes and two study visits each lasting approximately 6 - 8 hours. The investigators are looking for healthy, non-smoking male and female volunteers between the ages of 18 - 65, with no medical history of diabetics, heart, lung, kidney, stomach, or liver disease.

The initial screening visit will determine subject' eligibility through height, weight and waist circumference measurements, blood glucose (finger prick) test and a fasting screening blood draw. There will be no compensation for the screening visit, other than transportation costs.

If subject qualify, subject will continue to the two study visits. Each visit will require subject to have blood drawn several times during subject' study visit (total amount of blood equal to approximately 1 ½ tablespoons). To make this process more tolerable, a registered nurse will place a catheter (similar to what happens when you give blood) into subject's vein for ease in drawing blood. After the catheter placement and the first blood draw, subject will be asked to eat the test meal (tomato or non-tomato meal) and then subject will continue to have blood taken at specific time points for the next 6 hours. The investigators will also do an ultrasound on subject's arm to measure blood flow both before eating and midway through the 6 - hour study visit. The investigators will ask that subject not consume tomatoes or tomato products during the course of the study and record all food and beverages consumed on certain days.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* Between ages of 18-65
* BMI between 19 and 24 and hsCRP < 1mg/L
* BMI between 25 and 35 and hsCRP > 2.5mg/L
* No clinical evidence of cardiovascular, respiratory, renal, GI or hepatic disease

Exclusion Criteria:

* Pregnant and/or lactating
* allergies or intolerances to foods consumed in the study
* fasting blood glucose > 110mg/dL
* taking OTC antioxidant supplements, prescription meds that may interfere with study endpoints
* unusual dietary habits
* actively trying to lose or gain weight
* addicted to drugs or alcohol
* medically documented psychiatric or neurological disturbances
* smoker (past smoker allowed if cessation > 2 years)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, MS, PhD, Principal Investigator — Clinical Nutrition Research Center, Illinois Institute of Technology; Indika Edirisinghe, PhD, Principal Investigator — Clinical Nutrition Research Center, Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Burton-Freeman B, Talbot J, Park E, Krishnankutty S, Edirisinghe I. Protective activity of processed tomato products on postprandial oxidation and inflammation: a clinical trial in healthy weight men and women. Mol Nutr Food Res. 2012 Apr;56(4):622-31. doi: 10.1002/mnfr.201100649. Epub 2012 Feb 14. PMID 22331646

RESULTS

PARTICIPANT FLOW:
Groups:
- Tomato First Then Non-tomato: Tomato :High fat meal with tomato
- Non-tomato First Then Tomato: Non-tomato :High fat meal with non-tomato
Period: Overall Study
Arm/Group | Tomato First Then Non-tomato | Non-tomato First Then Tomato
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of twenty five subjects completed the crossover study (n = 12 females, n = 13 males).
Groups:
- Tomato First Then Non-tomato: tomato High fat test meal
  Tomato products: tomato with High fat test meal
- Non-tomato First Then Tomato: Non-tomato high fat test meal
  Non-tomato test meal: non-tomato with High fat test meal
- Total: Total of all reporting groups
Arm/Group | Tomato First Then Non-tomato | Non-tomato First Then Tomato | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.9 (5) | 28.7 (10.7) | 27 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 5 | 8 | 13

OUTCOME MEASURES:

1. Primary Outcome: IL-6 Concentrations
Time Frame: 6 hour postprandial study
Population: Analysis was per-protocol (tomato vs Non-tomato) and no imputations were given for any missing values; missing values treated as a missing.
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Groups:
- Tomato: High fat tomato test meal
  Tomato products: High fat tomato test meal
- Non-tomato: Non-tomato high fat test meal
  Non-tomato test meal: High fat non-tomato test meal
Arm/Group | Tomato | Non-tomato
Number analyzed (Participants) | 25 | 25
pg/mL | 2.2 (0.27) | 2.6 (0.28)
Statistical Analysis 1: Comparison: Tomato vs Non-tomato; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

ADVERSE EVENTS:
Arm/Group | Tomato | Non-tomato
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
Acute study; Chronic effect should be investigated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes